CLINICAL TRIAL: NCT00618787
Title: Prospective Randomized Double Blind Clinical Trial of Polyhexamethylene Biguanide Impregnated Foam Dressing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tyco Healthcare Group (Industry)
Responsible Party: Tonya Eggleston, RN, MPH, Study Director, Tyco Healthcare Group
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 360.18
Record Dates: First submitted 2008-01-10; First posted 2008-02-20 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Device: COPA AMD (note: name is not an acronym)
- Arm 2 (Active Comparator)
  Interventions: Device: COPA (note: name is not an acronym)

INTERVENTIONS:
Device: COPA AMD (note: name is not an acronym) — Foam dressing impregnated with Polyhexamethylene Biguanide
  Arms: Arm 1
Device: COPA (note: name is not an acronym) — Regular foam dressing without PHMB
  Arms: Arm 2

SUMMARY:
This is a multi-center, prospective, randomized, double blind, pilot clinical trial of subjects with chronic wounds. The purpose of this study is to compare the efficacy of COPA AMD PHMB Impregnated foam dressing compared to regular foam dressing in subjects with chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* subject is 18 to 85 years of age inclusive
* subject has a foot ulcer
* subject has a leg ulcer
* subject has an open wound of at 1.0 cm (2)
* subject has one of the following: Palpable pulse, ABI > 0.56 or toe pressure > 50 mmHg
* subject or legally authorized rep is able to understand and willing to give written informed consent

Exclusion Criteria:

* subject has an allergy to Chlorhexidine Gluconate (CHG)
* subject has open wounds that in the opinion of the Principal Investigator do not have the ability to heal
* subject has current malignant disease or history of malignant disease in past 5 years
* subject has inability to comply with the study protocol and procedures
* subjects who require use of topical agents other than the impregnated or regular foam dressings dressings

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Gary Sibbald, MD, Principal Investigator — Community Dermatology and Wound Healing Clinic, Women's College Hospital- Dermatology Daycare & Wound Healing Clinic
Locations (2):
- Canada (2):
  - Community Dermatology and Wound Healing Clinic, Mississauga, Ontario
  - Women's College Hospital; Dermatology Daycare & Wound Healing Clinic, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first study subject was randomized on March 5, 2008 and the last subject visit was conducted on February 18, 2009. Subjects were screened for eligibility, consented, enrolled and randomized at two participating wound care clinics.
Groups:
- COPA AMD: Foam dressing impregnated with Polyhexamethylene Biguanide
- COPA: Regular foam dressing without Polyhexamethylene Biguanide
Period: Overall Study
Arm/Group | COPA AMD | COPA
Started | 22 | 23
Completed | 19 | 21
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COPA AMD | COPA | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 21 | 37
  >=65 years | 6 | 2 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (15.28) | 55.1 (11.01) | 55.8 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Signs of Critical Colonization, Deep Infection, and Wound Healing Between the Two Groups
Time Frame: 5 weeks
Reporting Status: Not Posted

2. Secondary Outcome: Pain
Time Frame: 5 weeks
Reporting Status: Not Posted

3. Primary Outcome: Percentage Change in Wound Surface Area (cm2) at Week 4 Compared to Week 0.
Description: At each study visit, the subject's wound surface area was measured by longest length times widest width at right angles (LxW=cm2). Compiled data were analyzed to determine the median percentage decrease in wound surface area between groups and between study visits. Results report the median percentage decrease of the wound surface area as measured by cm2, comparing wound surface area at Week 4 to Week 0.
Time Frame: Weeks 0 and 4
Population: Per protocol
Measure: Median (Full Range); unit: Percentage change
Arm/Group | COPA AMD | COPA
Number analyzed (Participants) | 19 | 21
Percentage change | 34.9 [-74.8 to 94.7] | 27.8 [-167 to 97.6]

ADVERSE EVENTS:
Time Frame: One year
Description: Adverse events were assessed during each study visit (bi-weekly clinic visits) and as they occurred (e.g., adverse event is reported to the research team by subject, family member or other healthcare professional). Assessment type was a protocol specific coding system based on anticipated adverse events and physiological systems.
Arm/Group | COPA AMD | COPA
Serious Adverse Events (participants affected / at risk) | 0/22 | 2/23
Other Adverse Events (participants affected / at risk) | 5/22 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPA AMD (N=22) | COPA (N=23)
cardiac stent implanted (Cardiac disorders) | 0 (0) | 1 (1)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPA AMD (N=22) | COPA (N=23)
Head, eyes, ears, nose and throat (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Skin/Dermatologic (not including study wound) (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (3)
Wound Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Endocrine, metabolic and nutritional (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Allergic and immunologic (Endocrine disorders) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Digestive/Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urogenital (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematopoietic/Lymphatic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No